CLINICAL TRIAL: NCT07139886
Title: Phase 2b Multi-center Clinical Trials to Clarify the Efficacy and Adaptation Target of DA9601 in Patients With Acute and Chronic Gastritis, and to Determine the Optimal Clinical Dosage and Administration.
Brief Title: A Study to Evaluate the Safety and Efficacy of DA9601 for Acute and Chronic Gastritis and to Determine the Optimal Clinical Dosage and Administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA9601_GAS_IIb
Record Dates: First submitted 2025-08-18; First posted 2025-08-24 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Acute Gastritis; Chronic Gastritis
MeSH Terms: interventions — DA 9601

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): administered 2 tablets of placebo three times daily for two weeks
  Interventions: Drug: Stillen® Tab Placebo
- DA-9601(Stillen®) 180mg (Experimental): administered 1 tablet of placebo and 1 tablet of DA-9601(Stillen®) three times daily for two weeks
  Interventions: Drug: Stillen® Tab; Drug: Stillen® Tab Placebo
- DA-9601(Stillen®) 360mg (Experimental): administered 2 tablets of DA-9601(Stillen®) three times daily for two weeks
  Interventions: Drug: Stillen® Tab

INTERVENTIONS:
Drug: Stillen® Tab — Oral administration 3 times per day (in-between meals and before sleep) for 2 weeks
  Arms: DA-9601(Stillen®) 180mg; DA-9601(Stillen®) 360mg
Drug: Stillen® Tab Placebo — Oral administration 3 times per day (in-between meals and before sleep) for 2 weeks
  Arms: DA-9601(Stillen®) 180mg; Placebo

SUMMARY:
This is a multicenter, placebo-controlled, randomized, double-blinded, paralleled group clinical study to evaluate the efficacy of 2-week treatment with DA-9601 tab in patients with acute or chronic gastritis. Subject will receive DA-9601 180mg, 360mg tab or Placebo., three times a day for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with acute gastritis and chronic gastritis by endoscopy; have gastric mucosal lesions such as erosion, bleeding, redness, swelling on the site; and have subjective and objective symptoms requiring medical treatment ② 18 years old or older, 75 years old or younger ③ Patients who have agreed with the terms of clinical trials

Exclusion Criteria:

* Patients with peptic ulcer (excluding scars) and reflux esophagitis

  * Patients who were administered with H2 antagonist, muscarine receptor antagonist or nonsteroidal anti-inflammatory drug within 2 weeks prior to the start of the trial

    * Patients using protective agent enhancers at the start of the trial ④ Patients with recurrence observed during maintenance therapy at the start of the trial

      * Patients with a history of gastrectomy

        * Patients with severe disorders of the liver, kidneys, heart, lungs, blood, etc. ⑦ Patients with duodenal ulcer ⑧ Patients with gastrointestinal malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 1997-03-14 (Actual); Primary Completion 1999-07-08 (Actual); Study Completion 1999-07-08 (Actual)

PRIMARY OUTCOMES:
Change in Subjective and Objective Symptoms, Gastroscopy, Overall Improvement, Effectiveness grade | 2 weeks
  evaluated in 5 levels of "Significant improvement • Moderate improvement • Mild improvement • No improvement • Exacerbation"

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University Medical Center, Division of Gastroenterology, Suwon, Gyeonggi-do, South Korea